CLINICAL TRIAL: NCT03961880
Title: Impact of Recurrence Score on Adjuvant Treatment Decisions and Tumor Cell Dissemination in Estrogen-receptor Positive and HER2 Negative Patients With Early Breast Cancer
Brief Title: Impact of Recurrence Score on Adjuvant Treatment Decisions in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: IRMA
Record Dates: First submitted 2019-05-14; First posted 2019-05-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
IRMA is a Prospective, monocenter, non-interventional investigator initiated (IIT) registry that aims to investigate the use of the CE-marked OncotypeDX and its impact on adjuvant therapy recommendations in the clinical routine. Additionally, the proportion of patients with low, intermediate and high RS in predefined clinical subgroups will be determined. To evaluate the impact of the RS on tumor cell dissemination, these subgroups also include DTC-negative versus DTC-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* women ≥ 18 years of age
* histologically proven unilateral primary non-metastatic invasive breast cancer
* ER-/ or PR- positive and HER2-negative
* N0-N1 (0-3 involved lymph-nodes). The nodal status may be evaluated clinically.
* surgery or planed surgery at the Department of women's health, Tuebingen
* written informed consent into IRMA

Exclusion Criteria:

* ER-negative
* HER2-positive
* > 3 involved lymph-nodes
* bilateral breast cancer
* preexisting cancer disease within the last 10 years
* preexisting invasive ipsi- or contralateral breast cancer (non-invasive ipsi- or contralateral breast cancer is not regarded as an exclusion criteria)
* primary systemic therapy
* locally advanced, inoperable or metastatic breast cancer
* pregnant or lactating patients
* inadequate general condition (not fit for chemotherapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the influence of the 21-gene Recurrence-Score (RS) on adjuvant therapy recommendation | 1 year
  The Recurrence Score is a continuous score that provides an individual estimate of the 10 year risk of distant recurrence and predicts the likelihood of benefit from chemotherapy. The quantitative nature of PCR allows for a continuous score as opposed to a binary result (low vs. high only). Oncotype DX test results assign a Recurrence Score - a number between 0 and 100 - to the early-stage breast cancer or DCIS.
  Recurrence Score lower than 18: The cancer has a low risk of recurrence. The benefit of chemotherapy is likely to be small and will not outweigh the risks of side effects.
  Recurrence Score of 18 up to and including 30: The cancer has an intermediate risk of recurrence. It's unclear whether the benefits of chemotherapy outweigh the risks of side effects.
  Recurrence Score greater than or equal to 31: The cancer has a high risk of recurrence, and the benefits of chemotherapy are likely to be greater than the risks of side effects.

SECONDARY OUTCOMES:
Evaluation of the association of the RS with tumor cell dissemination into bone marrow | 1 year
  Bone marrow sampling is performed during primary surgery as part of the clinical routine. The presence of disseminated tumor cells (DTC status) is evaluated by immunostaining.
Correlation of the RS with age | 1 year
  age in years
Correlation of the RS with tumor nodal status | 1 year
Correlation of the RS with tumor grading | 1 year
Correlation of the RS with proliferation marker Ki-67 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Women's Health, Tübingen, Baden-Wurttemberg, Germany